CLINICAL TRIAL: NCT03678805
Title: Evaluation of the Efficiency of Minimally-invasive Surgically-assisted Withdrawal of Palatally Impacted Maxillary Canines in Terms of Movement Velocity and Dento-alveolar Changes: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Surgical Interventions to Assist Orthodontic Movement of Impacted Maxillary Canines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-19 -2018
Record Dates: First submitted 2018-09-17; First posted 2018-09-20 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Impaction of Tooth
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceleration (Experimental): The impacted canines will undergo acceleration by corticotomy accompanied with traditional traction techniques.
  Interventions: Procedure: Corticotomy
- Traditional Traction (Active Comparator): Traditional traction will be employed in this group of patients with impacted canines.
  Traditional withdrawal techniques will be used.
  Interventions: Procedure: Traditional withdrawal techniques

INTERVENTIONS:
Procedure: Corticotomy — Perforations in the areas close to the impacted canines will be performed in order to accelerate tooth movement.
  Arms: Acceleration
Procedure: Traditional withdrawal techniques — The impacted canines will be withdrawn using elastic modules.
  Arms: Traditional Traction

SUMMARY:
Impacted canine causes many problems for patients, such as absorption and damages to the adjacent teeth roots, as well as aesthetic problems. Correction of this problem requires a lengthy time. Therefore, many methods have been suggested to accelerate the movement of impacted canines with the help of surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Palatal or Mid-alveolar impacted canine.
2. There is no previous orthodontic treatment.
3. Healthy periodontal tissues and good oral health (i.e., Plaque Index is less or equal to 1 according to Loe and Silness(1963)).
4. No consumption of any drug that may interfere with the tooth movement (Cortisone, NSAIDs, …).
5. Mild or no crowding in the upper jaw.
6. No history of previous trauma to the maxillofacial region or surgical interventions.

Exclusion Criteria:

1. Any systemic diseases that would affect tooth movement
2. Antidepressant prevents oral surgery
3. Any congenital syndromes or cleft lip and palate cases
4. Bad oral health
5. Previous orthodontic treatment

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Duration of Canine Traction | The required time (in days) to achieve complete alignment of the impacted canine will be calculated which is expected to occur within 10-12 months in the traditional group and 7-8 months in the accelerated group
  The time required in days will be calculated from the beginning of canine traction till the end of canine alignment in its place in the dental arch.
Change in Canine Location in the Axial View | T1: one day before the beginning of treatment; T2: at the end of the traction stage which is expected to occur within 10-12 months in the traditional group and 7-8 months in the accelerated group.
  The distance between the cusp tip of the impacted canine to the palatal mid-line in the axial view using cone-beam computed tomography (CBCT) imaging.
Change in Canine Inclination in the Coronal View | T1: one day before the beginning of treatment; T2: at the end of the traction stage which is expected to occur within 10-12 months in the traditional group and 7-8 months in the accelerated group.
  The mesiodistal inclination of the impacted canine will be calculated which is the angle between the long axis of the impacted canine and the mid-sagittal plane in the coronal view of the cone-beam computed tomography (CBCT) imaging.
Change in the Canine Inclination in the Sagittal View | T1: one day before the beginning of treatment; T2: at the end of the traction stage which is expected to occur within 10-12 months in the traditional group and 7-8 months in the accelerated group.
  The labiopalatal inclination of the impacted canine: will be calculated which is the angle between the long axis of the impacted canine and a line perpendicular to the horizontal plane in the sagittal view of the cone-beam computed tomography (CBCT) imaging.
Change in the 3D Canine Location | T1: one day before the beginning of treatment; T2: at the end of the traction stage which is expected to occur within 10-12 months in the traditional group and 7-8 months in the accelerated group.
  The vertical distance from the cusp tip of the impacted canine to the upper occlusion plane is measured using the 3D volumetric rendered model of the cone-beam computed tomography (CBCT) imaging.
Relation to adjacent teeth | Just one day before the beginning of treatment
  The contact between the impacted canine and the central and/or the lateral incisor will be evaluated by looking at the shortest distance between the impacted canine crown and the adjacent incisors' roots This will be done using sequential axial views on the cone-beam computed tomography (CBCT) imaging.
Change in the Absorption to the adjacent roots | T1: one day before the beginning of treatment; T2: at the end of the traction stage which is expected to occur within 10-12 months in the traditional group and 7-8 months in the accelerated group.
  Absorption of adjacent roots will be evaluated as follows:
  In the axial views: an estimation of root damage will be taken into account and will be combined with an estimation of the vertical root damage using 3D volumetric rendered models and then will be classified into one of the four categories Class I: cementum involvement only and located at the apical third of the root Class II: involvement reaching the dentin but vertically less than one-third of the root length.
  Class III: involvement reaching the dentin and partially the pulp but still vertically less than one-third of the root length.
  Class IV: involvement reaching the root pulp and damaging more than one third of the root length vertically.

CONTACTS AND LOCATIONS:
Overall Officials: Mahran Mousa, DDS MSc, Principal Investigator — PhD Student in Orthodontics, University of Damascus Dental School, Damascus; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Associate Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria; Omar Heshmeh, DDS MSc PhD, Study Director — Associate Professor of Oral and Maxillofacial Surgery, Oral and Maxillofacial Surgery Department, University of Damascus Dental School, Damascus, SYRIA
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer TJ. Orthodontic treatment acceleration with corticotomy-assisted exposure of palatally impacted canines. Angle Orthod. 2007 May;77(3):417-20. doi: 10.2319/0003-3219(2007)077[0417:OTAWCE]2.0.CO;2. PMID 17465647
- [Background] Sukh R, Singh GP, Tandon P. Interdisciplinary approach for the management of bilaterally impacted maxillary canines. Contemp Clin Dent. 2014 Oct;5(4):539-44. doi: 10.4103/0976-237X.142828. PMID 25395776
- [Background] Shastri D, Nagar A, Tandon P. Alignment of palatally impacted canine with open window technique and modified K-9 spring. Contemp Clin Dent. 2014 Apr;5(2):272-4. doi: 10.4103/0976-237X.132362. PMID 24963263
- [Background] Baccetti T, Leonardi M, Armi P. A randomized clinical study of two interceptive approaches to palatally displaced canines. Eur J Orthod. 2008 Aug;30(4):381-5. doi: 10.1093/ejo/cjn023. Epub 2008 Jun 3. PMID 18524761
- [Background] Leonardi M, Armi P, Franchi L, Baccetti T. Two interceptive approaches to palatally displaced canines: a prospective longitudinal study. Angle Orthod. 2004 Oct;74(5):581-6. doi: 10.1043/0003-3219(2004)0742.0.CO;2. PMID 15529490
- [Background] Sebaoun JD, Surmenian J, Dibart S. [Accelerated orthodontic treatment with piezocision: a mini-invasive alternative to conventional corticotomies]. Orthod Fr. 2011 Dec;82(4):311-9. doi: 10.1051/orthodfr/2011142. Epub 2011 Nov 23. French. PMID 22105680
- [Background] Walker L, Enciso R, Mah J. Three-dimensional localization of maxillary canines with cone-beam computed tomography. Am J Orthod Dentofacial Orthop. 2005 Oct;128(4):418-23. doi: 10.1016/j.ajodo.2004.04.033. PMID 16214621
- [Background] Smailiene D, Kavaliauskiene A, Pacauskiene I, Zasciurinskiene E, Bjerklin K. Palatally impacted maxillary canines: choice of surgical-orthodontic treatment method does not influence post-treatment periodontal status. A controlled prospective study. Eur J Orthod. 2013 Dec;35(6):803-10. doi: 10.1093/ejo/cjs102. Epub 2013 Jan 24. PMID 23349422
- [Background] Alqerban A, Jacobs R, van Keirsbilck PJ, Aly M, Swinnen S, Fieuws S, Willems G. The effect of using CBCT in the diagnosis of canine impaction and its impact on the orthodontic treatment outcome. J Orthod Sci. 2014 Apr;3(2):34-40. doi: 10.4103/2278-0203.132911. PMID 24987661